CLINICAL TRIAL: NCT05656872
Title: A Comparative Study Between Transverse Abdominis Plane Block Versus Ilioinguinal-iliohypogastric Block For Postoperative Analgesia Following Open Abdominal Hysterectomy : A Randomized Controlled Trial
Brief Title: Transverse Abdominis Plane Block Versus Ilioinguinal-iliohypogastric Block For Analgesia Following Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Youssef Ollaek, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS-617-2021
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block (Active Comparator): Transversus abdominus plane (TAP) block will be used as postoperative analgesia
  Interventions: Procedure: Transverse Abdominis Plane Block
- IIIH Block (Active Comparator): Ilioinguinal-iliohypogastric (IIIH) block will be used as postoperative analgesia
  Interventions: Procedure: Ilioinguinal-iliohypogastric block

INTERVENTIONS:
Procedure: Transverse Abdominis Plane Block — Group T, will be performed in a supine position after skin sterilization, a linear high-frequency transducer Siemens acuson x300 3-5 MHZ will be placed in the transverse plane to the lateral abdominal wall in the mid-axillary line, between the lower costal margin and iliac crest. The abdominal wall muscles (external oblique, internal oblique, and transversus abdominis) will be visualized. A blunt tip,20-gauge, short bevel needle(Pajunk Sonoplex, Germany) will be inserted in-plane and advanced anterior to posterior under continuous visualization until the tip reaches between the internal oblique and the transversus abdominis muscle. After negative aspiration, 20 mL of bupivacaine 0.25%, lidocaine 1% will be injected. Separation of the internal oblique and transversus abdominis with a distinct pocket of local anesthetic in-between will be observed. The procedure will be repeated following the same steps on the other side.
  Arms: TAP Block
Procedure: Ilioinguinal-iliohypogastric block — Group I, will receive an Ultrasound-guided IIIH block that will be performed in a supine position after skin sterilization, a linear high-frequency transducer Siemens acuson x300 3-5 MHZ will be placed on the line between the anterior superior iliac spine and the umbilicus, where 3 layers of muscles (extra-abdominal oblique, intra-abdominal oblique, and transverse abdominis) will be visible on the inner side of the anterior superior iliac spine.A blunt tip,20-gauge, short bevel needle(Pajunk Sonoplex, Germany) will be inserted in-plane and advanced anterior to posterior under continuous visualization until the tip reaches between the internal oblique and the transversus abdominis muscle next to the iliohypogastric/ilioinguinal nerve. After negative aspiration, 20 mL of bupivacaine 0.25%, lidocaine 1% will be injected. The procedure will be repeated following the same steps on the other side.
  Arms: IIIH Block

SUMMARY:
The investigators hypothesis that ilioinguinal iliohypogastric nerves block could provide a potent modality of postoperative pain control as compared to Transverse Abdominis Plane block in open abdominal hysterectomy

DETAILED DESCRIPTION:
Aim of the work

the aim of the study is to compare between the analgesic effect of Transverse Abdominis Plane Block and Ilioinguinal-iliohypogastric block following open abdominal hysterectomy Objectives

* to compare between the analgesic effect of Transverse Abdominis Plane Block and Ilioinguinal-iliohypogastric block For Postoperative Analgesia following open abdominal hysterectomy
* to measure the incidence of complications following both blocks as hematoma, block failure, infection at injection site

Sample size:

Our primary outcome is the time to first rescue analgesia request. In a previous study, the meantime to first rescue analgesia was 10.58 ± 2.35 hours (6). The investigators calculated a sample size that could detect a mean difference of 20% between both study groups. MedCalc Software version 14 (MedCalc Software bvba, Ostend, Belgium) was used to calculate the sample size.38 patients( 19 patients per group) at least were estimated to have a study power of 80% and an alpha error of 0.05. This number will be increased to 42 patients (21 patients per group) to compensate for possible dropouts.

Sample size calculation was performed guided by the power of 80%, confidence level of 95%.

Statistical analysis:

For data analysis, the Statistical Package for Social Science (SPSS) software, version 26 for Microsoft Windows (SPSS Inc., Chicago, IL, USA) will be used. The Chi-squared test will be used to examine categorical data, which will be given as frequency (percent). The Shapiro-Wilk test will be used to verify for normality in continuous data, and the results will be provided as mean (standard deviation) or median (interquartile range) as appropriate. Depending on the data's normality, the unpaired t-test or the Mann Whitney test will be used to assess it. Repeated measures will be examined using analysis of variance (ANOVA), with posthoc pairwise comparisons using the Bonferroni tests. A P value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adult patients (18-65 years)
* ASA I-II
* Scheduled for elective open TAH

Exclusion Criteria:

* Patient refusal
* Any known allergy to local anesthetic
* Patients with neurological, psychological disorders or those lacking cooperation
* Patients with anatomic abnormalities at site of injection, skin lesions or wounds at site of proposed needle insertion.
* Patients with bleeding disorders defined as (INR >2) and/ or (platelet count <100,000/µL)
* Patients with hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia request | Immediatly post operative for 24 hours
  Time to first rescue analgesia request

SECONDARY OUTCOMES:
Total nalbuphine consumption in each block (mg) | Immediate 24 hours post-operative
  Total nalbuphine consumption in each block (mg)
VAS score | Immediate post-operative period every 5 minutes for the first 30 minutes , 2 hours, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours.
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10 centimeters line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Intraoperative hemodynamics | At baseline, 5 minutes after intubation, every 10 minutes till the end of the surgery, immediately after extubation, 5 minutes after extubation, and every 10 minutes in PACU for 30 minutes till the discharge of the patient
  Heart Rate (HR) beats/min. Mean Arterial Blood Pressure (mg)
Incidence of postoperative nausea and vomiting | Immediate 24 hours post-operative
  Incidence of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Ollaek, MD, Principal Investigator — Department of Anesthesia, Surgical ICU and Pain Management
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Cairo University, Cairo
  - Mohamed Ollaek, Cairo

IPD SHARING:
Plan to Share IPD: No